CLINICAL TRIAL: NCT05437783
Title: Influence of Ethnicity and ABCB1 Gene Polymorphism on the Pharmacokinetics of Azithromycin in Healthy Bangladeshi Volunteers: A Preliminary Study.
Brief Title: Influence of Ethnicity and ABCB1 Gene Polymorphism on the Pharmacokinetics of Azithromycin in Healthy Bangladeshi Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Zakia Sultana Ahmed, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BSMMU/2022/933
Record Dates: First submitted 2022-06-18; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Comparative Bioavailability Study
Keywords: Azithromycin; ABCB1 Gene; Pharmacokinetics; Single Nucleotide Polymorphism
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Bangladeshi Bangalee volunteers (Active Comparator): Bangladeshi bangalee participants will be fasting overnight for 10 h, all subjects will receive a single oral dose of 500mg of azithromycin with 250 ml of water. Drug intake will be ensured by direct supervision. Standardized meals will be served 4 and 10 h after dosing. Venous blood sample will be collected at multiple timepoints beginning before drug administration (0h) and containing at timepoints 1.0,2.0,3.0,4.0,6.0,8.0,12.0,24.0,48.0 and 72.0h post dosing. Two ml peripheral blood will be collected from each subject for genetic study.
  Interventions: Drug: Azithromycin Dihydrate
- Healthy Bangladeshi minor ethnics volunteers (Active Comparator): Bangladeshi minor ethnics participants will be fasting overnight for 10 h, all subjects will receive a single oral dose of 500mg of azithromycin with 250 ml of water. Drug intake will be ensured by direct supervision. Standardized meals will be served 4 and 10 h after dosing. Venous blood sample will be collected at multiple timepoints beginning before drug administration (0h) and containing at timepoints 1.0,2.0,3.0,4.0,6.0,8.0,12.0,24.0,48.0 and 72.0h post dosing. Two ml peripheral blood will be collected from each subject for genetic study.
  Interventions: Drug: Azithromycin Dihydrate

INTERVENTIONS:
Drug: Azithromycin Dihydrate — exclusively hospitalized at Bandarban Sadar hospital, Bandarban, Bangladesh. Participants will be fasting overnight for 10 h, all subjects will receive a single oral dose of 500mg of azithromycin with 250 ml of water. Drug intake will be ensured by direct supervision. Standardized meals will be served 4 and 10 h after dosing. Venous blood sample will be collected at multiple timepoints beginning before drug administration (0h) and containing at timepoints 1.0,2.0,3.0,4.0,6.0,8.0,12.0,24.0,48.0 and 72.0h post dosing. Two ml peripheral blood will be collected from each subject for genetic study.
  Other Names: Azithromycin

SUMMARY:
It is well recognized that different patients respond in different ways to the same medication. These differences are often greater among members of a population than they are within the same person at different times (or between monozygotic twins). The existence of large population differences with small interpatient variability is consistent with inheritance as a determinant of drug response; it is estimated that genetics can account for 20 to 95 percent of variability in drug disposition and effects. Azithromycin is frequently used worldwide irrespective of gender or ethnic populations therefore, to investigate the impact of gender and ABCB1 gene polymorphism holds clinical significance. As a correlation between azithromycin high plasma level and cardiac arrhythmia also exists . If we can prove the variation of pharmacokinetics of azithromycin due to ethnic differences and ABCB1 polymorphism dose adjustment can be done.

No relevant study regarding this has been done before in Bangladesh. Therefore, this preliminary study would be of great benefit to formulate the individualized doses regiment design which may improve the efficacy of drug while reducing adverse reaction. At the same time, Genotyping may prove an essential tool for individualized treatment by optimizing the drug dosage for an individual's genetic variability. Further study regarding pharmacogenetics of various drugs may be possible in our country in the future .The present study design to investigate the influence of ethnic difference and gene polymorphism on the pharmacokinetics of azithromycin in Bangladeshi Bangalee and Bangladeshi minor ethnic volunteers.

DETAILED DESCRIPTION:
Individual variation in drug response is a major problem in clinical practices and drug development which ranges from therapeutic failure to adverse drug reaction as drug reaction in multidrug therapy. Pharmacogenetic is relevant in this aspect and mainly concern with the study of genetic variation, which influence individuals' responses to drug. Again, polymorphism (variation) in the genes which are involved in encoding drug metabolizing enzymes, transporters of drug and ion channels can play role in the adverse drug reaction in an individual or can interfere with the therapeutic efficacy. For this reason, now-a-days concept of drug treatment is changed from 'right drug for the right person' to 'right dose for the right person at right time'. The human multidrug resistance gene ATP-binding cassette (ABCB1) codes for P-glycoprotein(P-gp), an important membrane-bound efflux transporter known to confer anticancer drug resistance as well as affect the pharmacokinetics of many drugs and xenobiotics. A number of single nucleotide polymorphisms (SNPs) have been identified throughout the ABCB1 gene that may have effect on P-gp expression levels and functions. Some studies shown an association between ABCB1 gene polymorphism on the pharmacokinetics of azithromycin. Genetic studies to explain this topic is uncommon. On this context, this proposed preliminary study is therefore to investigate the impact of ethnic difference and ABCB1 gene polymorphism on the pharmacokinetics of azithromycin among Bangladeshi people. This study will be a single dose open level comparative pharmacokinetic study, which will be conducted in the department of Pharmacology, BSMMU with the collaboration of Department of Anatomy, BSMMU and Bandarban Sadar Hospital, Bandarban. In this study healthy Bangladeshi volunteers will be divided into two arms-Bangladeshi Bengalese and Bangladeshi minor ethnics residing Chittagong Hill Tracts area, a total of 30 healthy volunteers of aged 20-25 will be provided 500mg oral azithromycin tablet and blood samples will be collected before drug administration (oh) and continuing at time points ,0.5 1.0, 2.0, 3.0, 4.0, 6.0, 8.0, 12.0, 24.0, 48.0, 72.0 h post dosing.2ml peripheral blood will be collected from each subject to determine the ABC1B gene polymorphism. This proposed study we would attempt to establish a High-Performance liquid Chromatography (HPLC) method to determine the azithromycin in plasma, in order to evaluate the bioavailability of azithromycin. Specific Genotypic polymorphism ABCB1 gene would be determine by Polymerase Chain Reaction-Restriction fragmentation Length Polymorphism Analysis (RFLP-PCR). After estimation of azithromycin and genotyping ABCB1 gene polymorphism, statistical analysis will be done to compare those values.

ELIGIBILITY:
Inclusion Criteria: 1. Healthy Bangladeshi male and female subjects, between the ages of 20 and 25 years. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate (PR) measurement, 12-lead ECG, routine laboratory tests (Blood chemistry, hematology and urine analysis).

2. BMI of 18 to 28 kg/m2; and a total body weight ≥50 kg for males and ≥45 kg for females.

3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

4. Subjects must be the residence of Chittagong Hill Tracts by birth.

-

Exclusion Criteria:

1. Liver cirrhosis.
2. Chronic renal failure. .
3. History of gastrectomy.
4. History of drug abuse within the past 5 years.
5. Treatment with an investigational drug within 3 months preceding the first dose of investigational product.
6. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the subject's eligibility.
7. Screening supine 12-lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS complex >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
8. Female subjects who are breastfeeding or with positive pregnancy test at Screening and during the study period.
9. Use of prescription or nonprescription drugs, dietary supplements and herbal medicines within 14 days prior to Screening.
10. Blood donation (excluding plasma donations) or loss of blood of approximately 450 mL or more within 3 months prior to Screening.

111. History of hypersensitivity to azithromycin or any components of its formulation.

112. Use of special diet (including dragon fruit, grape fruit juice, mango, citrus, etc.), strenuous activities or other factors that may affect the disposition of the study medication within 14 days prior to Screening.

13. Use of chocolate, food or beverages containing caffeine or xanthine within 48 hours prior to dosing.

14. Use of products containing alcohol within 48 hours prior to dosing. 15. History of HIV, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HCVAb..

16. Schizophrenia or other psychiatric illness..

-

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | [pre -dose(baseline) and day 1, day 2, day 3 post dose as designed time intervals.
  Maximum observed plasma concentration of Azithromycin
AUC0-t | [pre -dose(baseline) and day 1, day 2, day 3 post dose as designed time intervals.
  Area under the plasma concentration-time curve from time 0 to time t
AUC0-inf | [pre -dose(baseline) and day 1, day 2, day 3 post dose as designed time intervals.
  Area under the plasma concentration-time curve from time 0 to infinity

SECONDARY OUTCOMES:
Tmax | [pre -dose(baseline) and day 1, day 2, day 3 post dose as designed time intervals.
  Time of maximum plasma concentration of azithromycin
t1/2 | [pre -dose(baseline) and day 1, day 2, day 3 post dose as designed time intervals.
  Elimination half life
Identification of genotypic of polymorphism of the gene ABCB1coding for P-gp. | 2.o hours of post dosing.
  To investigate the existence of a relation between single nucleotide polymorphism of ABCB1 and plasma concentration of azithromycin

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh